CLINICAL TRIAL: NCT04688814
Title: (SEQ Block): Single Puncture Combined Lumbar Erector Spinae Plane Block and Quadratus Lumborum Block for Perioperative Analgesia in Acetabular Surgeries
Brief Title: SEQ Block for Perioperative Analgesia in Acetabular Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, moustafa abdelaziz, Professor of Anaesthesia and Surgical Intensive Care, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0304884
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Anesthesia, Local; Nerve Pain; Pain, Postoperative; Acetabular Fracture
MeSH Terms: conditions — Neuralgia; Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine Group (Active Comparator): Patients will receive GA and analgesia will be based on opioids mainly intravenous morphine. Intravenous morphine in a dose of 0.05 mg/kg will be given as a rescue analgesic when the VAS ≥4 postoperatively for 24 hours
  Interventions: Drug: Morphine Sulfate
- SEQ group (Experimental): Patients will receive ultrasound guided SEQ block preoperatively before the induction of general anaesthesia. Twenty five ml of 0.25 % bupivacaine will be given in the QL plane and 25 ml of the same concentration will be given in the erector spine plane
  Interventions: Procedure: Single puncture combined lumbar erector spinae plane block and quadrates lumborum block

INTERVENTIONS:
Procedure: Single puncture combined lumbar erector spinae plane block and quadrates lumborum block — Patients will lay laterally with the fracture side independent, a curvilinear transducer will be placed in a parasagittal plane 3-4 cm lateral to the lumbar spinous process of L4.The probe is shifted slowly to the lateral side till the transverse processes disappear. After subcutaneous local infiltration with lidocaine 1% at the cephalic end of the probe, the block needle is advanced through the erector spinae and QL muscles, until it pierces the epimysium of the QL muscle. LA is injected anterior to the QL, between the QL and psoas muscles.
  Then the caudal end of the probe is rotated slowly medially towards lumbar spine till the transverse process of L4 appears in the ultrasound image. The needle is withdrawn to subcutaneous tissue, then advanced in plane towards transverse process of L4. After contacting it, LA is deposited between transverse process and overlying ESM.
  Other Names: SEQ group
  Arms: SEQ group
Drug: Morphine Sulfate — Patients will receive GA and analgesia will be based on opioids mainly intravenous morphine
  Other Names: MOR group
  Arms: Morphine Group

SUMMARY:
The study will evaluate ultrasound guided SEQ block: single puncture combined lumbar erector spinae plane block and paraspinous sagittal shift (PSSS) quadratus lumborum block when compared with conventional intravenous morphine analgesia in patients undergoing posterior column acetabular fracture surgery

DETAILED DESCRIPTION:
Introduction: Acetabular fractures represent relatively infrequent traumatic injuries that can lead to a progressive impairment of hip articular function. Surgical treatment of these fractures may require extensive surgical dissections and frequently is associated with significant postoperative pain, delay in rehabilitation, and prolonged hospital stay. Innervation of the acetabular region is mainly provided by branches of lumbar and sacral plexuses, in addition to dorsal rami of lumbar nerve roots supplying the tissues to be dissected during posterior approach for acetabular fractures. Investigators suggest a novel approach for combined lumbar erector spinae plane block and PSSS quadratus lumborum block for perioperative analgesia in hip/acetabular surgeries using a single puncture technique (SEQ block).

Aim of the study: The primary aim of this study is to compare the total postoperative opioid (morphine) consumption after posterior column acetabular surgery when providing ultrasound guided SEQ block: single puncture combined lumbar erector spinae plane block and paraspinous sagittal shift (PSSS) quadratus lumborum block versus conventional intravenous morphine analgesia.

The secondary aims of this study are; intraoperative and postoperative hemodynamics; Mean arterial blood pressure (MAP) and heart rate (HR), resting visual analogue scale (VAS), dynamic VAS and postoperative complications.

Methods: After obtaining approval from Alexandria university ethics committee, this study will be carried out starting from December 2020 for 1 year in Alexandria university hospital on 52 American Society of Anesthesiologists (ASA) physical status I-III patients scheduled for unilateral posterior wall/column acetabular fractures surgery using posterior approach. The exclusion criteria will include; Body mass index (BMI) > 35 kg/m2, pre-existing neurological deficit, spine deformity, pregnancy/lactation, significant renal or hepatic impairment, known contraindications to peripheral nerve block (coagulopathy or infection at the site of injection), or chronic opioid users/abusers.

Patients will be divided randomly by closed envelope method into 2 groups. Group SEQ; patients will receive ultrasound guided SEQ block preoperatively before the induction of general anaesthesia (GA).

Group MOR; patients will receive GA and analgesia will be based on opioids mainly intravenous morphine.

Upon arrival to the operating room (OR), a multichannel monitor will be attached to patients, followed by the administration of 2 mg midazolam IV after securing an IV cannula.

Group SEQ: SEQ block is a combination of paraspinous sagittal shift (PSSS) quadratus lumborum (QL) block and erector spinae plane block (ESPB). Before the induction of GA in group SEQ, patients will lay laterally on the healthy side with the fracture side independent, a curvilinear ultrasound transducer (2-5 MHz) (Sonosite, M-turbo, Bothell, WA, USA) will be placed in a parasagittal plane 3-4 cm lateral to the lumbar spinous process of L4 (which is almost opposite to the iliac crest), producing a longitudinal scan of the lumbar paravertebral region, thus identifying the transverse processes of L3 and L4 with psoas muscle (PM) in-between and erector spinae muscle (ESM) posteriorly (superficial to transverse processes), the probe is shifted slowly to the lateral side till the transverse processes disappear and quadratus lumborum (QL) muscle is evident in its long axis attached caudally to the iliac crest with a characteristic sonographic image of three muscle layers appearing from posterior to anterior as : ESM, QL, and PM muscles respectively. Here, anterior layer of thoracolumbar fascia (ATLF) - which is considered as a continuation of fascia transversalis - is seen separating PM and QL muscles.

After subcutaneous local infiltration with lidocaine 1% at the cephalic end of the probe, the block needle is advanced in a cephalo-caudal direction, through the erector spinae and QL muscles, until it pierces the epimysium of the QL muscle. Local anaesthetic (LA) is injected anterior to the QL, observing it's spread in a caudal direction towards the iliac crest between the QL and psoas muscles.

Then the caudal end of the probe is rotated slowly medially towards lumbar spine till the hypoechoic shadow of transverse process of L4 appears in the ultrasound image. The needle is withdrawn to subcutaneous tissue, then advanced in plane towards transverse process of L4. After contacting it, LA is deposited in the plane between transverse process and overlying ESM. Total volume of LA used will be 50 ml of 0.25 % bupivacaine, 25 ml for each injection.

While, in group MOR; no block will be given. General anaesthesia will be induced with propofol 2 mg/kg, atracurium 0.5 mg/kg, and fentanyl 1µg/kg, followed by endotracheal intubation, anaesthesia will be maintained by isoflurane 1 Minimum Alveolar Concentration (MAC) in 100% oxygen. Multimodal analgesia protocol will be provided including intravenous dexamethasone 8 mg, paracetamol 1 gm, and ketorolac 60 mg. Increments of 0.5 µg/kg of fentanyl will be given intraoperatively if there is an increase in HR/MAP above 20% of the basal value.

Postoperatively, multimodal analgesia regimen will be continued in the form of paracetamol 1 g /8 hours and ketorolac 30 mg /8 hours intravenously for 24 hours. Intravenous morphine in a dose of 0.05 mg/kg will be given as a rescue analgesic when the VAS ≥4.

Measurements:

1. HR and MAP will be recorded preoperatively (baseline), every 30 minutes during the surgery, and every hour postoperatively for the first 4 hours, then every 4 hours for the remaining 24 hour postoperative follow up.
2. Resting VAS every hour for the first 4 hours, then every 4 hours for the remaining 24 hour postoperative follow up.
3. Dynamic VAS every hour for the first 4 hours, then every 4 hours for the remaining 24 hour postoperative follow up.
4. Total analgesic requirement (intraoperative fentanyl and postoperative morphine).
5. Postoperative complications (block or opioid related complications).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III patients
* Unilateral posterior wall/column acetabular fractures surgery using posterior approach

Exclusion Criteria:

* BMI > 35 kg/m2
* Pre-existing neurological deficit
* Spine deformity
* Pregnancy/lactation
* Significant renal impairment
* Significant Hepatic impairment
* Known contraindications to peripheral nerve block (coagulopathy or infection at the site of injection)
* Chronic opioid users/abusers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Total postoperative morphine consumption | 24 hours postoperatively
  Compare the total postoperative opioid (morphine) consumption after posterior column acetabular surgery when providing ultrasound guided SEQ block: single puncture combined lumbar erector spinae plane block and paraspinous sagittal shift (PSSS) quadratus lumborum block versus conventional intravenous morphine analgesia. Morphine 0.05 mg/kg will be given intravenously when VAS score is ≥ 4. The total postoperative morphine consumption in milligrams will be recorded.

SECONDARY OUTCOMES:
Heart rate (HR) | 24 hours
  HR (beats/minute) will be recorded preoperatively (baseline), every 30 minutes during the surgery, and every hour postoperatively for the first 4 hours, then every 4 hours for the remaining 24 hour postoperative follow up. Hemodynamic measurement will be done using multichannel Mindray monitor MEC-1000, mindray Ltd, Shenzhen, China
Mean arterial blood pressure (MABP) | 24 hours
  MABP (mmHg) will be recorded preoperatively (baseline), every 30 minutes during the surgery, and every hour postoperatively for the first 4 hours, then every 4 hours for the remaining 24 hour postoperative follow up. Hemodynamic measurement will be done using multichannel Mindray monitor MEC-1000, mindray Ltd, Shenzhen, China
Resting and dynamic visual analogue score | 24 hours
  Every patient will be asked postoperatively according to a visual analogue scale (VAS) score from 0 -10 about his experience with pain. Zero is equal to the best pain relief and 10 is referring to the worst pain experience. This will be also asked about during active movement of the hip joint and will be interpreted as the dynamic pain score. This will be done every hour during the 1st 4 postoperative hours and every 4 hours later for the rest 24 hour follow up period.
Postoperative complications | 24 hours
  Block or opioid related complications Nausea and vomiting: Incidence and frequency Urine retention: Incidence and frequency Any manifestation of nerve injury like the presence of paresthesia: Incidence and frequency

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa A Moustafa, Professor, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request
Supporting Information: Study Protocol
Time Frame: Data will become available after 1 year for one year
Access Criteria: Via mail of the principal investigator

REFERENCES:
- [Background] Chelly JE, Casati A, Al-Samsam T, Coupe K, Criswell A, Tucker J. Continuous lumbar plexus block for acute postoperative pain management after open reduction and internal fixation of acetabular fractures. J Orthop Trauma. 2003 May;17(5):362-7. doi: 10.1097/00005131-200305000-00007. PMID 12759641
- Available data/document: Study Protocol — http://www.med.alexu.edu.eg

DOCUMENTS (1):
  • Study Protocol (2020-12-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04688814/Prot_000.pdf